CLINICAL TRIAL: NCT00259064
Title: A Phase II Multicentre Randomised, Parallel Group, Double-Blind, Placebo-Controlled Study of ZD1839 (IRESSATM) (250MG Tablet) Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Chemotherapy-Naive Patients With Advanced (Stage IIIB or IV) Non-Small Cell Lung Cancer (NSCLC) and Poor Performance Status
Brief Title: Iressa v BSC (Best Supportive Care) in First Line NSCLC
Acronym: INSTEP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0711; D7913C00711
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: NSCLC
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Gefitinib (Experimental): ZD1839 + BSC (best supportive care)
  Interventions: Drug: Gefitinib
- Placebo (Placebo Comparator): Placebo + BSC (best supportive care)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gefitinib
  Arms: Gefitinib
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if the addition of Iressa to Best Supportive Care treatment will increase the progression free survival of chemo-naïve, poor performance status patients, with stage IIIB or IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* NSCLC - locally advanced (Stage IIIB) or metastatic (stage IV) disease, not amenable to curative surgery or radiotherapy
* Not suitable for chemotherapy
* WHO Performance status 2 or 3

Exclusion Criteria:

* Newly diagnosed CNS mets
* Less than 4 weeks since completion of radiotherapy or persistence of any radiotherapy related toxicity
* Other co-existing malignancies
* ALT/AST greater than 5 x upper limit of normal
* ANC less than 1.0 x 109/L or platelets less than 100 x 109/L

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To compare Iressa v best supportive care in terms of progression free survival | Progression-free survival

SECONDARY OUTCOMES:
To compare Iressa v best supportive care in terms of objective tumour response rate | Overall objective tumour response rate (CR and PR) according to the RECIST criteria
To compare Iressa v best supportive care in terms of overall survival | Time to death
To compare Iressa v best supportive care in terms of quality of life | Improvement in patient-reported functionality as measured by trial outcome index, comprised of the physical and functional well being sections and LCS of FACT-L and quality of life measured by the FACT-L total score
To compare Iressa v best supportive care in terms of tolerability | Adverse event profile (type, frequency and severity of adverse events); laboratory parameters and vital signs

OTHER OUTCOMES:
To investigate the correlation of the expression of biomarkers in tumour tissue obtained prior to gefitinib therapy with gefitinib clinical efficacy and to determine a set of biomarkers to enable patient selection for therapy. | Efficacy (objective response rate and progression free survival), toxicity, EGFR signalling pathways markers, RNA expression profile, gene polymorphisms of pre specified germline and tumour genes, DNA methylation, plasma and urine proteomics
To compare gefitinib + BSC versus Placebo + BSC in terms of Health Resource Utilisation | The use of selected items of resource and concomitant medications including: number of in patient days, number of out patient visits, number of invasive procedures, pallative radiotherapy, concomitant medications.
To compare gefitinib + BSC versus Placebo + BSC in terms of changes in pain and fatigue | Changes in pain and fatigue as measured by the single items from the FACT-L physical well being domain.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (36):
- Australia (7):
  - Research Site, Bedford Park
  - Research Site, Chermside
  - Research Site, Concord
  - Research Site, Melbourne
  - Research Site, Newcastle
  - Research Site, Prahran
  - Research Site, Randwick
- Canada (18):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
- Research Site, Nová Ves pod Pleší, Czechia
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, The Hague
  - Research Site, Zutphen
- United Kingdom (5):
  - Research Site, Abergavenny
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, Wolverhampton

REFERENCES:
- See also: CSR-1839IL-0711.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1550&filename=CSR-1839IL-0711.pdf